CLINICAL TRIAL: NCT02266264
Title: Hyperglycemia and Effects of Daily 100 Milligrams Versus 200 Milligrams of Hydrocortisone Therapy in Patients With Septic Shock: A Double-Blind Randomized Controlled Trial
Brief Title: Hyperglycemia and Effects of Daily 100 mg Versus 200 mg of Hydrocortisone Therapy in Patients With Septic Shock
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Srinakharinwirot University (Other)
Responsible Party: Principal Investigator, Kanchana Ngaosuwan, Doctor, Srinakharinwirot University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MED-R2R-200
Record Dates: First submitted 2014-10-10; First posted 2014-10-17 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 100 milligrams of hydrocortisone (Experimental): 100 milligrams per day of hydrocortisone is the starting dosage.
  Interventions: Drug: Hydrocortisone
- 200 milligrams of hydrocortisone (Active Comparator): 200 milligrams per day of hydrocortisone is the starting dosage.
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — Subjects will be divided into two groups by randomization. The intervention-group will be received 100 milligrams per day of hydrocortisone and the control-group will be received 200 milligrams per day of hydrocortisone in the first three days after enrollment.
  Other Names: solu cortef

SUMMARY:
The purpose of this study is to compare hyperglycemia and other effects, include 28-day mortality and time to reversal of shock between 100 milligrams and 200 milligrams of hydrocortisone as initial dosage in patients with septic shock.

DETAILED DESCRIPTION:
The intervention group will be received 100 milligrams per day of hydrocortisone on the first three day the taper off, whereas the control group will be received 200 milligrams per day of hydrocortisone on the first three day the taper off. Hyperglycemia rate will be monitored every 6 hours after hydrocortisone is started until 24 hours after it is stopped.

Also, 28-day mortality will be follow after hydrocortisone is started.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock
* Adequate fluid resuscitation and vasopressor therapy are unable to maintain hemodynamic stability

Exclusion Criteria:

* Receive systemic steroid in past 3 months
* Established adrenal insufficiency
* Currently used in chemotherapy or immunosuppressive agents
* Radiotherapy currently received
* Known HIV infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Hyperglycemia | two years
  Proportion of hyperglycemic patients

SECONDARY OUTCOMES:
28-day mortality | two years
  The number of the patients who died before or at 28 days after enrollment.
Time to shock reversal | two years
  The dates when vasopressors can be stopped.

CONTACTS AND LOCATIONS:
Overall Officials: Kanchana Ngaosuwan, Master, Principal Investigator — Department of Medicine, Faculty of Medicine, Srinakharinwirot University
Locations (1):
- Department of Medicine, Faculty of Medicine, Srinakharinwirot University, Ongkharak, Changwat Nakhon Nayok, Thailand